CLINICAL TRIAL: NCT05296369
Title: Randomized Controlled Clinical Study of Folic Acid Treatment of Radiation Esophagitis After Chemoradiation in Lung Cancer
Brief Title: Folic Acid Interferes With Radiation Esophagitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guizhou Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GZMU-FA
Record Dates: First submitted 2022-03-04; First posted 2022-03-25 (Actual); Last update posted 2022-03-25 (Actual); Status verified 2022-03

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Folic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Folic acid intervention
  Interventions: Drug: Folic acid
- Routine (No Intervention): Routine treatment intervention

INTERVENTIONS:
Drug: Folic acid — Folic acid was added during the period prior to concurrent chemoradiotherapy
  Arms: Experimental

SUMMARY:
This randomized study compared the incidence and severity of radiation esophagitis with folic acid and with conventional symptomatic treatment.

DETAILED DESCRIPTION:
By prospective randomized controlled study, this study research plans to recruit with diagnosis of lung cancer patients, according to whether there is drug intervention were divided into treatment group and control group, compared two groups of acute radiation esophagitis in the before and after the intervention, extent of occurrence of folic acid and clinical curative effect, so as to verify whether folic acid can be used as an intervention in the treatment of radioactive esophagitis, To explore the safety of folic acid in the treatment of radioactive esophagitis and explore the standardized treatment of radioactive esophagitis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with malignant lung cancer (incluedig Non-small cell lung cancer, small cell lung cancer) diagnosed by histopathology or cytology.
2. TNM Stage N2~N3 (IASLC International TNM staging standard for Lung Cancer, 8th edition) was indicated by radiotherapy and the patients were treated for the first time.
3. Aged between 18 and 75 years old,no limit on the gender.
4. ECOG≤2 or KPS≥70.
5. No contraindication of Concurrent chemoradiotherapy.
6. Patients without important organ dysfunction,hematology: it is within the normal range according to the standards of each laboratory; Cardiac function: normal range; Liver function: normal range; Renal function: normal range; Pulmonary function: FEV1 > 50%, mild to moderate impairment of pulmonary function.
7. Patients with good compliance to treatment received and follow-up.

Exclusion Criteria:

1. Prior to treatment, there were other esophageal diseases, such as gastrointestinal ulcer, reflux esophagitis, cardia relaxation.
2. Patients with severe nutritional anemia prior to treatment.
3. The IV stage patients with uncontrolled malignant pleural effusion,with diffuse liver or lung metastasis which lead to liver or pulmonary dysfunction.
4. Patients with severe heart, lung or kidney diseass,such as uncontrolled hypertension, diabetes, unstable angina, a history of myocardial infarction or heart failure, or uncontrolled arrhythmias; There is clearly clinically diagnosed heart valve disease; The active phase of a bacterial, fungal, or viral infection; Mental disorders; Severely impaired lung function.
5. A history of previous tumors complicated with other malignant tumors.
6. The pregnant or breast-feeding patients.
7. Patients with mental and neurological diseases.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival(PFS) | up to 12 months
  PFS is defined as the duration of time from start of treatment to time of progression or death, whichever occurs first.

SECONDARY OUTCOMES:
Severity of radiation esophagitis | day 1 up to 4 weeks after the end of treatment
  A modified NCI-CTC score (the sum of dysphagia pain score and dysphagia pain score) was used to evaluate the occurrence of radioactive esophagitis.
Number of participants with treatment-related adverse events as assessed by CTCAE v5.0 | day 1 up to 4 weeks after the end of treatment
  To assess and record nausea, vomiting, hematologic toxicity,radiation pneumonitis and other treantment complications by CTCAE v5.0.Hematotoxicity includes white blood cell count (The normal range count is 3.5 to 9.5×10^9/L), neutrophil count(The normal range count is 1.8 to 6.3×10^9/L), platelet count(The normal range count is 125 to 350×10^9/L), hemoglobin count(The normal range count is 115 to 175g/L),measuring creatinine value（The normal value of creatinine is 44to106μmol/L）, endogenous creatinine clearanceThe normal value of creatinine is 80 to120 mo/min）, bilirubin（Including total bilirubin, direct bilirubin and indirect bilirubin,), aspartate aminotransferase(AST, The normal value of AST is 13 to 40u/L)and alanine aminotransferase(ALT, The normal value of ALT is 7 to 50u/L).The severity of radiational pneumonitis can be evaluated by the Radiation Therapy Oncology Group（RTOG）morbidity grading criteria.

CONTACTS AND LOCATIONS:
Overall Officials: Bing Lu, MD, Principal Investigator — The affiliated Cancer Hospital of Guizhou Medical University
Locations (1):
- The Affiliated Cancer Hospital of Guizhou Medical University, Guiyang, Guizhou, China